CLINICAL TRIAL: NCT03796078
Title: Impact of Maxillomandibular Advancement Upon the Pharyngeal Airway Volume and the Apnea-hypopnea Index in the Treatment of Obstructive Sleep Apnea
Brief Title: Maxillomandibular Advancement in the Treatment of Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Dr. Federico Hernández-Alfaro MD, DDS, PhD, FEBOMS, Chief Oral and Maxillofacial Surgery Department, Centro Medico Teknon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSAS-OS
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: OSA; OSAS; Apnea, Obstructive Sleep; Orthognathic Surgery
Keywords: OSA; orthognathic surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Methylmalonic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bimaxillary surgery (MMA) (Active Comparator): Bimaxillary Orthognathic Surgery. MMA
  Interventions: Procedure: Maxillomandibular advancement
- monomaxillary surgery (Isolated MaxS) (Active Comparator): Monomaxillary surgery (Isolated MaxS)
  Interventions: Procedure: monomaxillary surgery (isolated MaxS)
- monomandibullary surgery (Isolated MandS) (Active Comparator): Monomandibular surgery (Isolated MandS)
  Interventions: Procedure: monomandibullary surgery (MandS)

INTERVENTIONS:
Procedure: Maxillomandibular advancement — Treatment: Mono or Bimaxillary Orthognathic Surgery. The surgery of Reposition of the jaws is carried out under general anesthesia using minimally invasive techniques, the patient is extubated After surgery, antibiotics are prescribed during admission, anti-inflammatories, antiemetics and a local cold mask is applied of closed circuit at 17ºCelsius. The patient is discharged at 24 h.
  Other Names: MMA (maxillomandibular advancement)
  Arms: Bimaxillary surgery (MMA)
Procedure: monomaxillary surgery (isolated MaxS) — Monomaxillary surgery (Isolated MaxS): The surgery of Reposition of the maxilla is carried out under general anesthesia using minimally invasive techniques, the patient is extubated After surgery, antibiotics are prescribed during admission, anti-inflammatories, antiemetics and a local cold mask is applied of closed circuit at 17ºCelsius. The patient is discharged at 24 h.
  Arms: monomaxillary surgery (Isolated MaxS)
Procedure: monomandibullary surgery (MandS) — Monomandibullary surgery (Isolated MandS): The surgery of Reposition of the maxilla is carried out under general anesthesia using minimally invasive techniques, the patient is extubated After surgery, antibiotics are prescribed during admission, anti-inflammatories, antiemetics and a local cold mask is applied of closed circuit at 17ºCelsius. The patient is discharged at 24 h.
  Arms: monomandibullary surgery (Isolated MandS)

SUMMARY:
ABSTRACT OBJECTIVES: To study the correlation between pharyngeal airway volume (PAV), the clinical indicators of obstructive sleep apnea (AHI, ESS), and the impact of orthognathic surgery on them.

METHODS: A prospective, descriptive, unicentric study carried out by a multidisciplinary team to evaluate the following parameters in patients undergoing orthognathic surgery at Maxillofacial institute Teknon medical center.

During the study period:

* Record of the type, magnitude and direction of surgical movements of the maxillofacial complex made during the surgery (Day 0-Month 1).
* Assessment of PAS/PAV stability (relapse) at short term (1 month).

  3D PAV assessment by cranial voxel-based superimposition protocol before and one month and 12 months after orthognathic surgery.
* Household polysomnography (PSG) registry/ apnea-hypopnea index (Day 0, Month 1 and Month 12). (AHI evaluation bu neurophysiologist)
* Assessment of the clinical indicators of obstructive sleep apnea at day 0, month 1 and month 12:, blood pressure (mm Hg) , and daytime hypersomnia test (Epworth sleepiness scale, ESS) (Day 0, Month 1 and Month 12).
* Record of body mass index (BMI) (cm/Kg2)

Main Objective:

• Evaluate the impact of orthognathic surgery (bimaxillary or monomaxillary) and its movements on the PAV and the clinical indicators of OSA.

Specific objectives:

• Interrelate the degree of dentofacial deformity with the IAH.

* Study the potential correlation between the volume of the VAS and the IAH.
* Correlate the type, direction and magnitude of the surgical movements of the maxillofacial complex with PAV/PAS increase Correlate the type, direction and magnitude of the surgical movements of the maxillofacial complex with the cure of OSA (household PSG AHI assessment) and the following clinical indicators of OSA: diurnal hypersomnia test (ESD, ESS).
* Evaluate negative effects of either maxillary or mandibular surgical movements in PAS/PAV increase and the cures of OSA.

Evaluate negative effects of either maxillary or mandibular surgical movements in the improvement of the clinical symptoms and the cure of OSA.

* To study the possible effect of surgical complications on PAS/PAV stability at long term and the clinical symptoms of OSA.
* Demonstrate that maxillomandibular surgery is a defined, predictable and a definitive cure for OSA.
* Demonstrate that skeletal, linear, and cross-sectional volume parameters remain stable at long-term.
* Demonstrate that AHI and OSA-related parameters stay stable at long term after mono- or bimaxillary surgery.

Hypothesis

* H1a: Maxillomandibular advancement (orthognathic surgery) does correlate with the volume of the upper airway, at both short or long term.
* H2a: Maxillomandibular advancement (orthognathic surgery) does correlate with the clinical indicators of obstructive sleep apnea, at both short or long term.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age who present any kind of dentofacial deformity candidates for orthognathic surgery treatment.
2. Growth of the maxillofacial complex completed.
3. Patients without uncontrolled cardio-pulmonary disease.
4. Patients willing to understand the procedures of the study and that agree to give their signed informed consent.
5. Patients who commit to perform the postoperative controls for at least one postoperative year.
6. Patients with a good general condition of health, confirmed by pre-operative study and assessment by Anaesthesiology (ASA).

Exclusion Criteria:

1. Patients with a clinical history in which any surgery would be contraindicated
2. Patients with any facial Syndromic malformation
3. Patients who have undergone chemotherapy or radiotherapy during the last 5 years, including area of head and neck.
4. Patients who refuse to accept the clinical conditions of the study and are not willing to sign the form corresponding informed consent.
5. Patients who are expected to lack adherence to follow-up or to the treatment.
6. Treatment with bisphosphonates or Denosumab (Prolia®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Upper airway volume change | Evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12).
  Evaluation of volume change of the pharyngeal airway before (Day 0) and month (Month 1) and 12 months (Month 12) comparing the three-dimensional measurements of maxillary /bimaxillary surgery by conical beam computed tomography superposition. Cubic millimeters (mm^3 will be used to evaluate this outcome)

SECONDARY OUTCOMES:
Pharyngeal airway space (amount of movement) | Evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12).
  Evaluation of the amount of movement (pharyngeal airway space increase) before (Day 0) and month (Month 1) and 12 months (Month 12) comparing the three-dimensional measurements of maxillary /bimaxillary surgery by conical beam computed tomography superposition. Millimeters will be used to determine this outcome
Direction of movement (advancement or setback) | Evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12).
  Evaluation of the direction of movement (advancement or setback) and its impact (negative/positive) in the total upper airway volume change, before (Day 0) and month (Month 1) and 12 months (Month 12) comparing the three-dimensional measurements of maxillary /bimaxillary surgery by conical beam computed tomography superposition. Millimetres will be used to determine this outcome.
Apnea-hypopnea index (AHI) assessment | Evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12).
  Evaluation of clinical indicators of obstructive sleep apnea: Apnea-hypopnea index by polysomnography evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12). AHI scale: Mild OSA 5-15/ moderate OSA: 15-30/ severe OSA: >30 events/hour. A higher score means a worse outcome.
Blood pressure changes | Evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12).
  Evaluation of clinical indicators of obstructive sleep apnea: blood pressure change evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12). Systolic and diastolic pressures will be both recorded. Mean cardiac frequency will be obtained.
  Evaluation of clinical indicators of obstructive sleep apnea: blood pressure change evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12). Systolic and diastolic pressures will be both recorded. Mean cardiac frequency will be obtained.
  Evaluation of clinical indicators of obstructive sleep apnea: blood pressure change evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12). Systolic and diastolic pressures will be both recorded. Mean cardiac frequency will be obtained. Assessed in mm Hg
Body mass index (BMI) | Evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12).
  Evaluation of Body mass index (e.g., weight in kilograms, height in m) change before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12). (e.g., weight and height will be combined to report BMI in kg/m^2).
Lowest oxygen saturation 90% (LSat 90%) | Evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12).
  Evaluation of clinical indicators of obstructive sleep apnea: lowest oxygen saturation (90%) change evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12).
Epworth sleepiness scale test (ESS) | Evaluated before surgery (Day 0), 1 month after surgery (Month 1) and 12 months after surgery (Month 12).
  The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness that is measured by use of a very short questionnaire. Used clinically to screen for the manifestations of the behavioral morbidity associated to obstructive sleep apnea, first used by Johns, 1991.
  The ESS asks people to rate, on a four-point scale, their usual chances of falling asleep in eight different situations. These must be answered beyond 4 punctuations ranges depending on: 0 = would never doze, 1 = slight chance of dozing, 2 = moderate chance of dozing or 3 = high chance of dozing. The total ESS score is the sum of item-scores and ranges between 0 and 24; the higher the score, the higher the person's level sleepines. A score of 10-12 is suggested as the cutoff among clinic populations being screened for a sleep disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Hernández-Alfaro, PhD, Study Chair — Institute of Maxillofacial Surgery, Teknon Medical Center; Adaia Valls-Ontañón, PhD, Principal Investigator — Institute of Maxillofacial Surgery, Teknon Medical Center
Locations (1):
- Institute of Maxillofacial Surgery, Teknon Medical Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giralt-Hernando M, Valls-Ontanon A, Guijarro-Martinez R, Masia-Gridilla J, Hernandez-Alfaro F. Impact of surgical maxillomandibular advancement upon pharyngeal airway volume and the apnoea-hypopnoea index in the treatment of obstructive sleep apnoea: systematic review and meta-analysis. BMJ Open Respir Res. 2019 Oct 9;6(1):e000402. doi: 10.1136/bmjresp-2019-000402. eCollection 2019. PMID 31673361
- [Background] Giralt-Hernando M, Valls-Ontanon A, Haas Junior OL, Masia-Gridilla J, Hernandez-Alfaro F. What are the Surgical Movements in Orthognathic Surgery That Most Affect the Upper Airways? A Three-Dimensional Analysis. J Oral Maxillofac Surg. 2021 Feb;79(2):450-462. doi: 10.1016/j.joms.2020.10.017. Epub 2020 Oct 15. PMID 33171114
- [Background] Hernandez-Alfaro F, Giralt-Hernando M, Brabyn PJ, Haas OL Jr, Valls-Ontanon A. Variation between natural head orientation and Frankfort horizontal planes in orthognathic surgery patients: 187 consecutive cases. Int J Oral Maxillofac Surg. 2021 Sep;50(9):1226-1232. doi: 10.1016/j.ijom.2021.02.011. Epub 2021 Feb 22. PMID 33632574

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03796078/Prot_SAP_002.pdf
  • Informed Consent Form (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03796078/ICF_003.pdf